CLINICAL TRIAL: NCT03626090
Title: Mesenchymal Stem Cell Therapy for Liver Cirrhosis: A Phase I/II Study
Brief Title: Mesenchymal Stem Cell Therapy for Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Med Pte. Ltd. (Industry)
Collaborators: Parkway Cancer Centre (Unknown); Asian American Liver Centre (Unknown); Desmond Wai Liver & Gastrointestinal Diseases Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-SM-L0001
Record Dates: First submitted 2018-07-26; First posted 2018-08-10 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
Keywords: Liver; Cirrhosis; Child B; Child C; Advance; Advanced; Singapore; MSC; Mesenchymal; Stem Cell; Cell Therapy; MSC Therapy; Treatment
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Intervention Model Description: As the primary objective of the study is to assess safety of MSC infusion, a single arm non-blinded study design has been adopted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A single dose of 0.5 to 1 x 10^6/kg autologous BM MSCs (Total volume: 30 - 50 ml) will be infused via peripheral venous access.
  Interventions: Biological: Autologous BM MSC

INTERVENTIONS:
Biological: Autologous BM MSC — A total of 100-200ml will be harvested from the subject, in either a single or multiple punctures. This will be processed for autologous MSC infusion.

SUMMARY:
MSCs have been studied for the treatment of liver diseases as well as non-liver diseases. MSCs have been successful in treating conditions like acute steroid-resistant GVHD in hematopoietic stem cell transplanted patients and also have shown to improve the MELD score in end-stage liver disease. There were no severe side effects observed in using autologous MSCs as a treatment option. The outcome of the studies done so far have been positive and it is encouraged to study the use of MSCs as cell therapy for treating liver diseases.

The estimated rate of cirrhosis in HBV patients in Singapore is about 1.6% per year, rate of hepatocellular carcinoma is about 0.8% per year overall and 3.0% per year in cirrhotic patients. Knowing that there are not many options currently available for Liver Cirrhosis patients and that they have a poor prognosis with an average life expectancy of < 12 months, this study uses autologous MSCs to treat Liver Cirrhosis patients in Singapore. The objective of the study is to demonstrate that autologous bone marrow is safe to be used in patients with liver cirrhosis as well as demonstrate that bone marrow MSC may improve liver function and prolong patient survival.

DETAILED DESCRIPTION:
Liver cirrhosis refers to extreme scarring of the liver, resulting in suboptimal function of the liver. It can result from a variety of causes, ranging from hepatitis B and C infection, excessive alcohol consumption, autoimmune causes, fatty liver and others. Irrespective of the cause, once the liver becomes cirrhotic, it is a downhill course.

Liver cirrhosis is irreversible and most patients will progressively worsen over time. Once liver cirrhosis has reached the stage of decompensation, that is, development of jaundice, ascites, variceal bleeding, hepatic encephalopathy and coagulopathy the two-year survival drops to about 50%.

The definitive treatment of decompensated cirrhosis is liver transplantation. While a liver transplantation is potentially curative, the high costs, lack of a donor, treatment-related mortality and the immunosuppression complications make this option possible only for a limited number of patients. The vast majority do not have an effective option at all, thus the need to develop alternative therapies. Various types of Stem Cells had been investigated as a regenerative therapy for liver cirrhosis. These stem cells include bone marrow mesenchymal stem cells (MSC), bone marrow mononuclear cells (MNC) and peripheral CD34 positive cells. Some early studies have shown encouraging results in patients who had autologous bone marrow stem cell transplantation. There was improved liver function in these patients with cirrhotic livers.

The sponsor is proposing a study to look into the role of MSC therapy for patients with liver cirrhosis in Singapore. This will be a Phase I/II study with the main emphasis on the safety profile first. The trial will be conducted in compliance with the protocol, GCP and local regulatory requirement(s).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the inclusive criteria to participate in the study:

1. with definite liver cirrhosis, irrespective of aetiology
2. must have Child's B or C stage
3. must have signed an informed consent form

Exclusion Criteria:

Subjects with any of the following criteria are regarded as an exclusion from the study and will not be permitted to participate:

1. age ≤21 years and >70 years old
2. with life expectancy of < 6 months
3. cancers and bone marrow malignancies
4. patients with an active infection or multiple infections
5. patients with uncontrolled hypertension and diabetes
6. immunosuppressed patients (IST must have stopped at least 4 weeks prior to trial enrolment)
7. patients who are HIV positive
8. patients who are pregnant or lactating

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-18 (Actual); Primary Completion 2021-10-22 (Estimated); Study Completion 2021-10-22 (Estimated)

PRIMARY OUTCOMES:
Clinical Examination | Up to 34 weeks
  To observe for the following:
  * absence of grade IV anaphylactic reactions (in reference to CTCAE 4.03)
  * absence of grade IV febrile reactions or septic/ infective complications (in reference to CTCAE 4.03).
MR Elastography | Up to 34 weeks
  To detect liver stiffness
The level of serum alanine aminotransferase (ALT) | Up to 34 weeks
  To ensure the absence of deterioration of liver function.
The level of glomerular filtration rate (GFR) | Up to 34 weeks
  To ensure the absence of deterioration of renal function.

SECONDARY OUTCOMES:
The level of serum prothrombin time (PT) | Up to 6 months, post-infusion
  To assess the efficacy of treatment
The level of serum total bilirubin (TB) | Up to 6 months, post-infusion
  To assess the efficacy of treatment
The level of serum albumin (ALB) | Up to 6 months, post-infusion
  To assess the efficacy of treatment
MELD Score | Up to 6 months, post-infusion
  To assess the efficacy of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Teo Cheng Peng, Principal Investigator — Parkway Cancer Centre; Wai Chun Tao, Desmond, Principal Investigator — Desmond Wai Liver & Gastrointestinal Diseases Centre; Lee Kang Hoe, Principal Investigator — Asian American Liver Centre
Locations (3):
- Singapore (3):
  - Asian American Liver Centre - Gleneagles Hospital (Annexe Block), Singapore
  - Parkway Cancer Centre - Gleneagles Hospital, Singapore
  - Desmond Wai Liver & Gastrointestinal Disease Centre - Mount Elizabeth Novena Specialist Centre, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poh Z, Goh BB, Chang PE, Tan CK. Rates of cirrhosis and hepatocellular carcinoma in chronic hepatitis B and the role of surveillance: a 10-year follow-up of 673 patients. Eur J Gastroenterol Hepatol. 2015 Jun;27(6):638-43. doi: 10.1097/MEG.0000000000000341. PMID 25831135
- [Background] Lyra AC, Soares MB, da Silva LF, Fortes MF, Silva AG, Mota AC, Oliveira SA, Braga EL, de Carvalho WA, Genser B, dos Santos RR, Lyra LG. Feasibility and safety of autologous bone marrow mononuclear cell transplantation in patients with advanced chronic liver disease. World J Gastroenterol. 2007 Feb 21;13(7):1067-73. doi: 10.3748/wjg.v13.i7.1067. PMID 17373741
- [Background] Terai S, Ishikawa T, Omori K, Aoyama K, Marumoto Y, Urata Y, Yokoyama Y, Uchida K, Yamasaki T, Fujii Y, Okita K, Sakaida I. Improved liver function in patients with liver cirrhosis after autologous bone marrow cell infusion therapy. Stem Cells. 2006 Oct;24(10):2292-8. doi: 10.1634/stemcells.2005-0542. Epub 2006 Jun 15. PMID 16778155
- [Background] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Background] Zhao DC, Lei JX, Chen R, Yu WH, Zhang XM, Li SN, Xiang P. Bone marrow-derived mesenchymal stem cells protect against experimental liver fibrosis in rats. World J Gastroenterol. 2005 Jun 14;11(22):3431-40. doi: 10.3748/wjg.v11.i22.3431. PMID 15948250
- [Background] Ortiz LA, Gambelli F, McBride C, Gaupp D, Baddoo M, Kaminski N, Phinney DG. Mesenchymal stem cell engraftment in lung is enhanced in response to bleomycin exposure and ameliorates its fibrotic effects. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8407-11. doi: 10.1073/pnas.1432929100. Epub 2003 Jun 18. PMID 12815096
- [Background] Meier RP, Muller YD, Morel P, Gonelle-Gispert C, Buhler LH. Transplantation of mesenchymal stem cells for the treatment of liver diseases, is there enough evidence? Stem Cell Res. 2013 Nov;11(3):1348-64. doi: 10.1016/j.scr.2013.08.011. Epub 2013 Aug 29. PMID 24090934
- [Background] Amorin B, Alegretti AP, Valim V, Pezzi A, Laureano AM, da Silva MA, Wieck A, Silla L. Mesenchymal stem cell therapy and acute graft-versus-host disease: a review. Hum Cell. 2014 Oct;27(4):137-50. doi: 10.1007/s13577-014-0095-x. Epub 2014 Jun 6. PMID 24903975
- [Background] Jacobs SA, Roobrouck VD, Verfaillie CM, Van Gool SW. Immunological characteristics of human mesenchymal stem cells and multipotent adult progenitor cells. Immunol Cell Biol. 2013 Jan;91(1):32-9. doi: 10.1038/icb.2012.64. PMID 23295415
- [Background] Uccelli A, Moretta L, Pistoia V. Mesenchymal stem cells in health and disease. Nat Rev Immunol. 2008 Sep;8(9):726-36. doi: 10.1038/nri2395. PMID 19172693
- [Background] Di Nicola M, Carlo-Stella C, Magni M, Milanesi M, Longoni PD, Matteucci P, Grisanti S, Gianni AM. Human bone marrow stromal cells suppress T-lymphocyte proliferation induced by cellular or nonspecific mitogenic stimuli. Blood. 2002 May 15;99(10):3838-43. doi: 10.1182/blood.v99.10.3838. PMID 11986244
- [Background] Krampera M, Glennie S, Dyson J, Scott D, Laylor R, Simpson E, Dazzi F. Bone marrow mesenchymal stem cells inhibit the response of naive and memory antigen-specific T cells to their cognate peptide. Blood. 2003 May 1;101(9):3722-9. doi: 10.1182/blood-2002-07-2104. Epub 2002 Dec 27. PMID 12506037
- [Background] Meisel R, Zibert A, Laryea M, Gobel U, Daubener W, Dilloo D. Human bone marrow stromal cells inhibit allogeneic T-cell responses by indoleamine 2,3-dioxygenase-mediated tryptophan degradation. Blood. 2004 Jun 15;103(12):4619-21. doi: 10.1182/blood-2003-11-3909. Epub 2004 Mar 4. PMID 15001472
- [Background] Suva D, Passweg J, Arnaudeau S, Hoffmeyer P, Kindler V. In vitro activated human T lymphocytes very efficiently attach to allogenic multipotent mesenchymal stromal cells and transmigrate under them. J Cell Physiol. 2008 Mar;214(3):588-94. doi: 10.1002/jcp.21244. PMID 17786951
- [Background] Kisseleva T, Cong M, Paik Y, Scholten D, Jiang C, Benner C, Iwaisako K, Moore-Morris T, Scott B, Tsukamoto H, Evans SM, Dillmann W, Glass CK, Brenner DA. Myofibroblasts revert to an inactive phenotype during regression of liver fibrosis. Proc Natl Acad Sci U S A. 2012 Jun 12;109(24):9448-53. doi: 10.1073/pnas.1201840109. Epub 2012 May 7. PMID 22566629
- [Background] Sheng H, Wang Y, Jin Y, Zhang Q, Zhang Y, Wang L, Shen B, Yin S, Liu W, Cui L, Li N. A critical role of IFNgamma in priming MSC-mediated suppression of T cell proliferation through up-regulation of B7-H1. Cell Res. 2008 Aug;18(8):846-57. doi: 10.1038/cr.2008.80. PMID 18607390
- [Background] Dmitrewski J, Olliff S, Buckels JA. Obstructive jaundice associated with polycystic liver disease. HPB Surg. 1996;10(2):117-20. doi: 10.1155/1996/83547. PMID 9184868
- [Background] Manousou P, Arvaniti V, Tsochatzis E, Isgro G, Jones K, Shirling G, Dhillon AP, O'Beirne J, Patch D, Burroughs AK. Primary biliary cirrhosis after liver transplantation: influence of immunosuppression and human leukocyte antigen locus disparity. Liver Transpl. 2010 Jan;16(1):64-73. doi: 10.1002/lt.21960. PMID 19866449
- [Background] Mohamadnejad M, Malekzadeh R, Nasseri-Moghaddam S, Hagh-Azali S, Rakhshani N, Tavangar SM, Sedaghat M, Alimohamadi SM. Impact of immunosuppressive treatment on liver fibrosis in autoimmune hepatitis. Dig Dis Sci. 2005 Mar;50(3):547-51. doi: 10.1007/s10620-005-2472-5. PMID 15810640
- [Background] Yang ZF, Ho DW, Ngai P, Lau CK, Zhao Y, Poon RT, Fan ST. Antiinflammatory properties of IL-10 rescue small-for-size liver grafts. Liver Transpl. 2007 Apr;13(4):558-65. doi: 10.1002/lt.21094. PMID 17394154
- [Background] Sgroi A, Gonelle-Gispert C, Morel P, Baertschiger RM, Niclauss N, Mentha G, Majno P, Serre-Beinier V, Buhler L. Interleukin-1 receptor antagonist modulates the early phase of liver regeneration after partial hepatectomy in mice. PLoS One. 2011;6(9):e25442. doi: 10.1371/journal.pone.0025442. Epub 2011 Sep 27. PMID 21980458
- [Background] Bartholomew A, Sturgeon C, Siatskas M, Ferrer K, McIntosh K, Patil S, Hardy W, Devine S, Ucker D, Deans R, Moseley A, Hoffman R. Mesenchymal stem cells suppress lymphocyte proliferation in vitro and prolong skin graft survival in vivo. Exp Hematol. 2002 Jan;30(1):42-8. doi: 10.1016/s0301-472x(01)00769-x. PMID 11823036
- [Background] Zappia E, Casazza S, Pedemonte E, Benvenuto F, Bonanni I, Gerdoni E, Giunti D, Ceravolo A, Cazzanti F, Frassoni F, Mancardi G, Uccelli A. Mesenchymal stem cells ameliorate experimental autoimmune encephalomyelitis inducing T-cell anergy. Blood. 2005 Sep 1;106(5):1755-61. doi: 10.1182/blood-2005-04-1496. Epub 2005 May 19. PMID 15905186
- [Background] Gerdoni E, Gallo B, Casazza S, Musio S, Bonanni I, Pedemonte E, Mantegazza R, Frassoni F, Mancardi G, Pedotti R, Uccelli A. Mesenchymal stem cells effectively modulate pathogenic immune response in experimental autoimmune encephalomyelitis. Ann Neurol. 2007 Mar;61(3):219-27. doi: 10.1002/ana.21076. PMID 17387730
- [Background] Augello A, Tasso R, Negrini SM, Cancedda R, Pennesi G. Cell therapy using allogeneic bone marrow mesenchymal stem cells prevents tissue damage in collagen-induced arthritis. Arthritis Rheum. 2007 Apr;56(4):1175-86. doi: 10.1002/art.22511. PMID 17393437
- [Background] Urban VS, Kiss J, Kovacs J, Gocza E, Vas V, Monostori E, Uher F. Mesenchymal stem cells cooperate with bone marrow cells in therapy of diabetes. Stem Cells. 2008 Jan;26(1):244-53. doi: 10.1634/stemcells.2007-0267. Epub 2007 Oct 11. PMID 17932424
- [Background] Lee KD, Kuo TK, Whang-Peng J, Chung YF, Lin CT, Chou SH, Chen JR, Chen YP, Lee OK. In vitro hepatic differentiation of human mesenchymal stem cells. Hepatology. 2004 Dec;40(6):1275-84. doi: 10.1002/hep.20469. PMID 15562440
- [Background] Li J, Tao R, Wu W, Cao H, Xin J, Li J, Guo J, Jiang L, Gao C, Demetriou AA, Farkas DL, Li L. 3D PLGA scaffolds improve differentiation and function of bone marrow mesenchymal stem cell-derived hepatocytes. Stem Cells Dev. 2010 Sep;19(9):1427-36. doi: 10.1089/scd.2009.0415. PMID 20055663
- [Background] Ong SY, Dai H, Leong KW. Inducing hepatic differentiation of human mesenchymal stem cells in pellet culture. Biomaterials. 2006 Aug;27(22):4087-97. doi: 10.1016/j.biomaterials.2006.03.022. Epub 2006 Apr 17. PMID 16616366
- [Background] Sato Y, Araki H, Kato J, Nakamura K, Kawano Y, Kobune M, Sato T, Miyanishi K, Takayama T, Takahashi M, Takimoto R, Iyama S, Matsunaga T, Ohtani S, Matsuura A, Hamada H, Niitsu Y. Human mesenchymal stem cells xenografted directly to rat liver are differentiated into human hepatocytes without fusion. Blood. 2005 Jul 15;106(2):756-63. doi: 10.1182/blood-2005-02-0572. Epub 2005 Apr 7. PMID 15817682
- [Background] Kuo TK, Hung SP, Chuang CH, Chen CT, Shih YR, Fang SC, Yang VW, Lee OK. Stem cell therapy for liver disease: parameters governing the success of using bone marrow mesenchymal stem cells. Gastroenterology. 2008 Jun;134(7):2111-21, 2121.e1-3. doi: 10.1053/j.gastro.2008.03.015. Epub 2008 Mar 12. PMID 18455168
- [Background] Seo MJ, Suh SY, Bae YC, Jung JS. Differentiation of human adipose stromal cells into hepatic lineage in vitro and in vivo. Biochem Biophys Res Commun. 2005 Mar 4;328(1):258-64. doi: 10.1016/j.bbrc.2004.12.158. PMID 15670778
- [Background] Chamberlain J, Yamagami T, Colletti E, Theise ND, Desai J, Frias A, Pixley J, Zanjani ED, Porada CD, Almeida-Porada G. Efficient generation of human hepatocytes by the intrahepatic delivery of clonal human mesenchymal stem cells in fetal sheep. Hepatology. 2007 Dec;46(6):1935-45. doi: 10.1002/hep.21899. PMID 17705296
- [Background] Natarajan A, Wagner B, Sibilia M. The EGF receptor is required for efficient liver regeneration. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17081-6. doi: 10.1073/pnas.0704126104. Epub 2007 Oct 16. PMID 17940036
- [Background] Parekkadan B, van Poll D, Megeed Z, Kobayashi N, Tilles AW, Berthiaume F, Yarmush ML. Immunomodulation of activated hepatic stellate cells by mesenchymal stem cells. Biochem Biophys Res Commun. 2007 Nov 16;363(2):247-52. doi: 10.1016/j.bbrc.2007.05.150. Epub 2007 May 30. PMID 17869217
- [Background] Ortiz LA, Dutreil M, Fattman C, Pandey AC, Torres G, Go K, Phinney DG. Interleukin 1 receptor antagonist mediates the antiinflammatory and antifibrotic effect of mesenchymal stem cells during lung injury. Proc Natl Acad Sci U S A. 2007 Jun 26;104(26):11002-7. doi: 10.1073/pnas.0704421104. Epub 2007 Jun 14. PMID 17569781
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Deeg HJ. How I treat refractory acute GVHD. Blood. 2007 May 15;109(10):4119-26. doi: 10.1182/blood-2006-12-041889. Epub 2007 Jan 18. PMID 17234737
- [Background] Tobin LM, Healy ME, English K, Mahon BP. Human mesenchymal stem cells suppress donor CD4(+) T cell proliferation and reduce pathology in a humanized mouse model of acute graft-versus-host disease. Clin Exp Immunol. 2013 May;172(2):333-48. doi: 10.1111/cei.12056. PMID 23574329
- [Background] Mohamadnejad M, Namiri M, Bagheri M, Hashemi SM, Ghanaati H, Zare Mehrjardi N, Kazemi Ashtiani S, Malekzadeh R, Baharvand H. Phase 1 human trial of autologous bone marrow-hematopoietic stem cell transplantation in patients with decompensated cirrhosis. World J Gastroenterol. 2007 Jun 28;13(24):3359-63. doi: 10.3748/wjg.v13.i24.3359. PMID 17659676
- [Background] Kharaziha P, Hellstrom PM, Noorinayer B, Farzaneh F, Aghajani K, Jafari F, Telkabadi M, Atashi A, Honardoost M, Zali MR, Soleimani M. Improvement of liver function in liver cirrhosis patients after autologous mesenchymal stem cell injection: a phase I-II clinical trial. Eur J Gastroenterol Hepatol. 2009 Oct;21(10):1199-205. doi: 10.1097/MEG.0b013e32832a1f6c. PMID 19455046
- [Background] Amer ME, El-Sayed SZ, El-Kheir WA, Gabr H, Gomaa AA, El-Noomani N, Hegazy M. Clinical and laboratory evaluation of patients with end-stage liver cell failure injected with bone marrow-derived hepatocyte-like cells. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):936-41. doi: 10.1097/MEG.0b013e3283488b00. PMID 21900788
- [Background] Zhang Z, Lin H, Shi M, Xu R, Fu J, Lv J, Chen L, Lv S, Li Y, Yu S, Geng H, Jin L, Lau GK, Wang FS. Human umbilical cord mesenchymal stem cells improve liver function and ascites in decompensated liver cirrhosis patients. J Gastroenterol Hepatol. 2012 Mar;27 Suppl 2:112-20. doi: 10.1111/j.1440-1746.2011.07024.x. PMID 22320928
- [Background] Gholamrezanezhad A, Mirpour S, Bagheri M, Mohamadnejad M, Alimoghaddam K, Abdolahzadeh L, Saghari M, Malekzadeh R. In vivo tracking of 111In-oxine labeled mesenchymal stem cells following infusion in patients with advanced cirrhosis. Nucl Med Biol. 2011 Oct;38(7):961-7. doi: 10.1016/j.nucmedbio.2011.03.008. Epub 2011 Jun 22. PMID 21810549
- [Background] Baertschiger RM, Serre-Beinier V, Morel P, Bosco D, Peyrou M, Clement S, Sgroi A, Kaelin A, Buhler LH, Gonelle-Gispert C. Fibrogenic potential of human multipotent mesenchymal stromal cells in injured liver. PLoS One. 2009 Aug 17;4(8):e6657. doi: 10.1371/journal.pone.0006657. PMID 19684854
- [Background] Forbes SJ, Russo FP, Rey V, Burra P, Rugge M, Wright NA, Alison MR. A significant proportion of myofibroblasts are of bone marrow origin in human liver fibrosis. Gastroenterology. 2004 Apr;126(4):955-63. doi: 10.1053/j.gastro.2004.02.025. PMID 15057733
- [Background] Casiraghi F, Remuzzi G, Abbate M, Perico N. Multipotent mesenchymal stromal cell therapy and risk of malignancies. Stem Cell Rev Rep. 2013 Feb;9(1):65-79. doi: 10.1007/s12015-011-9345-4. PMID 22237468
- [Background] Sundin M, Lindblom A, Orvell C, Barrett AJ, Sundberg B, Watz E, Wikman A, Broliden K, Le Blanc K. Persistence of human parvovirus B19 in multipotent mesenchymal stromal cells expressing the erythrocyte P antigen: implications for transplantation. Biol Blood Marrow Transplant. 2008 Oct;14(10):1172-1179. doi: 10.1016/j.bbmt.2008.08.003. PMID 18804048
- [Background] Sundin M, Orvell C, Rasmusson I, Sundberg B, Ringden O, Le Blanc K. Mesenchymal stem cells are susceptible to human herpesviruses, but viral DNA cannot be detected in the healthy seropositive individual. Bone Marrow Transplant. 2006 Jun;37(11):1051-9. doi: 10.1038/sj.bmt.1705368. PMID 16604097
- [Background] Zhou YF, Bosch-Marce M, Okuyama H, Krishnamachary B, Kimura H, Zhang L, Huso DL, Semenza GL. Spontaneous transformation of cultured mouse bone marrow-derived stromal cells. Cancer Res. 2006 Nov 15;66(22):10849-54. doi: 10.1158/0008-5472.CAN-06-2146. PMID 17108121
- [Background] Miura M, Miura Y, Padilla-Nash HM, Molinolo AA, Fu B, Patel V, Seo BM, Sonoyama W, Zheng JJ, Baker CC, Chen W, Ried T, Shi S. Accumulated chromosomal instability in murine bone marrow mesenchymal stem cells leads to malignant transformation. Stem Cells. 2006 Apr;24(4):1095-103. doi: 10.1634/stemcells.2005-0403. Epub 2005 Nov 10. PMID 16282438
- [Background] Dahl JA, Duggal S, Coulston N, Millar D, Melki J, Shahdadfar A, Brinchmann JE, Collas P. Genetic and epigenetic instability of human bone marrow mesenchymal stem cells expanded in autologous serum or fetal bovine serum. Int J Dev Biol. 2008;52(8):1033-42. doi: 10.1387/ijdb.082663jd. PMID 18956336
- [Background] Karnoub AE, Dash AB, Vo AP, Sullivan A, Brooks MW, Bell GW, Richardson AL, Polyak K, Tubo R, Weinberg RA. Mesenchymal stem cells within tumour stroma promote breast cancer metastasis. Nature. 2007 Oct 4;449(7162):557-63. doi: 10.1038/nature06188. PMID 17914389
- [Background] Rollin R, Alvarez-Lafuente R, Marco F, Jover JA, Hernandez-Garcia C, Rodriguez-Navas C, Lopez-Duran L, Fernandez-Gutierrez B. Human parvovirus B19, varicella zoster virus, and human herpesvirus-6 in mesenchymal stem cells of patients with osteoarthritis: analysis with quantitative real-time polymerase chain reaction. Osteoarthritis Cartilage. 2007 Apr;15(4):475-8. doi: 10.1016/j.joca.2006.11.007. Epub 2007 Jan 3. PMID 17207644
- [Background] Salama H, Zekri AR, Medhat E, Al Alim SA, Ahmed OS, Bahnassy AA, Lotfy MM, Ahmed R, Musa S. Peripheral vein infusion of autologous mesenchymal stem cells in Egyptian HCV-positive patients with end-stage liver disease. Stem Cell Res Ther. 2014 May 28;5(3):70. doi: 10.1186/scrt459. PMID 24886681
- [Background] Neagu M, Suciu E, Ordodi V, Unescu VP. Human Mesenchymal Stem Cells As Basic Tools for Tissue Engineering : Isolation and Culture. October. 2005;15(October):29-34.